CLINICAL TRIAL: NCT03930992
Title: Efficacy of 4 mg Zoledronic Acid Plus Colaren vs 4mg Zoledronic Acid + Conventional Treatment for Secondary Osteoporosis in HIV Positive and Negative Men
Brief Title: Efficacy of Zoledronic Acid + Colaren vs Zoledronic Acid + Conventional Treatment for Osteoporosis in HIV+ and HIV- Men
Acronym: OSZCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Luz Alicia González Hernández, Head of HIV Unit in Hospital Civil de Guadalajara, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSZCO
Record Dates: First submitted 2019-04-17; First posted 2019-04-29 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Secondary Osteoporosis
Keywords: 4 mg zoledronic acid; Colaren; HIV; Secondary Osteoporosis; Man
MeSH Terms: interventions — Seroconversion; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: Study type: Interventional, with four arms:
  1. arm: 4 mg zoledronic acid annually plus colaren ® in HIV-positive;
  2. arm: 4 mg zoledronic acid annually plus conventional treatment in HIV-positive;
  3. arm: 4 mg zoledronic acid annually plus colaren ® in HIV-negative;
  4. arm: 4 mg zoledronic acid annually plus conventional treatment in HIV-negative.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 Arm: Experimental (Experimental): Experimental: 4 mg zoledronic acid plus colaren ® This arm include: 20 man with HIV infection plus osteoporosis
  Interventions: Drug: Colaren in HIV positive
- 2 Arm: Active comparator (Active Comparator): Active comparator: 4mg zoledronic acid + standard treatment (or conventional treatment) This arm include: 20 man with HIV infection plus osteoporosis
  Interventions: Drug: standard treatment in HIV positive
- 3 Arm: Experimental (Experimental): Experimental: 4 mg zoledronic acid plus colaren ® This arm include: 20 man without HIV infection plus osteoporosis
  Interventions: Drug: Colaren in HIV negative
- 4 Arm: Active comparator (Active Comparator): Active comparator: 4mg zoledronic acid + standard treatment (or conventional treatment) This arm include: 20 man without HIV infection plus osteoporosis
  Interventions: Drug: standard treatment in HIV negative

INTERVENTIONS:
Drug: Colaren in HIV positive — 1 Arm (HIV+): will receive Zoledronic acid 4mg and colaren ® (vitamin D, magnesium, phosphate, calcium).
  Other Names: plus Zoledronic Acid 4 mg
  Arms: 1 Arm: Experimental
Drug: standard treatment in HIV positive — 2 Arm (HIV+): will receive Zoledronic acid 4mg and standard treatment (vitamin D and calcium carbonate)
  Other Names: plus Zoledronic Acid 4 mg
  Arms: 2 Arm: Active comparator
Drug: Colaren in HIV negative — 3 Arm (HIV-): will receive Zoledronic acid 4mg and colaren ® (vitamin D, magnesium, phosphate, calcium).
  Other Names: plus Zoledronic Acid 4 mg
  Arms: 3 Arm: Experimental
Drug: standard treatment in HIV negative — 4 Arm (HIV-): will receive Zoledronic acid 4mg and standard treatment (vitamin D and calcium carbonate)
  Other Names: plus Zoledronic Acid 4 mg
  Arms: 4 Arm: Active comparator

SUMMARY:
Clinical trial to assess the effectiveness of the supplement Colaren® associated with zoledronic acid 4mg/annually in the treatment of osteoporosis secondary, compared to standard treatment plus zoledronic acid 4mg/annually. The standard treatment will include 1gr of calcium/day and vitamin D supplement. In both cases, vitamin D levels will be determinated, which should remain at more than 30 ng/mL.

Including men with osteoporosis secondary to HIV and men with osteoporosis secondary to any other cause (HIV negative). Vitamin D levels, bone densitometry and markers of metabolism, bone formation and bone resorption will be assessment. The all parameters above will be assessed basally (before the start of treatment), after starting the treatment, an assessment will be made at 12 weeks where vitamin D levels and bone markers will be measured. Meanwhile, at week 24 assess only vitamin D levels; and finally, at week 52 all parameters mentioned above will be measured.

DETAILED DESCRIPTION:
This study is a clinical trial to assess the effectiveness of the supplement Colaren® associated with annually zoledronic acid 4mg, in the treatment of osteoporosis secondary or not to HIV infection, compared to standard treatment plus zoledronic acid 4mg/annually. The standard treatment will include 1gr of calcium/day and vitamin D supplement. In both cases, vitamin D levels will be evaluated, which should remain at more than 30 ng/mL.

Including men with osteoporosis secondary to HIV and men with osteoporosis secondary to any other cause (HIV negative). Vitamin D levels, bone densitometry and markers of metabolism, bone formation and bone resorption will be assessment. The all parameters above will be assessed basally (before the start of treatment), after starting the treatment, an assessment will be made at 12 weeks where vitamin D levels and bone markers will be measured. Meanwhile, at week 24 assess only vitamin D levels; and finally, at week 52 all parameters mentioned above will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adult males 18 to 65 years old.
* HIV diagnosis (HIV positive group) or negative HIV serology (HIV negative group).
* Patients receiving HAART and sustained virologic control for at least two years.
* Patients meeting diagnostic criteria for osteoporosis.
* Subjects willing to participate voluntarily in this study and give a written consent.
* Estimated glomerular filtration rate >60 mL/min (Using CKD-EPI formula).

Exclusion Criteria:

* Use of calcium, vitamin D or any other drug with bone activity during the last 90 days previous to the study.
* Use of herbs or herb products during the last 90 days previous to the study.
* Positive test for HCV or HBV.
* Patients who cannot be submitted to complete examination for variable analysis.
* Glomerular filtration rate <60 mL/minute.
* Active liver disease.
* Non-compliance to treatment (less than 90%).
* Patients who are not willing to continue participating.

Non-inclusion criteria:

* Female patients.
* Use of immunosuppressive o immunomodulatory treatment 90 days previous to selection.
* Use of prohibited drugs for the study like: antiestrogens, corticosteroids (doses greater than 7.5mg of prednisone/day) 90 days previous to selection.
* Use of hormone therapy.
* Patients with history or actual use of chemotherapy.
* Patients deprived of freedom or imprisoned patients with mental illnesses.
* Participant is part of another clinical trial or nutritional program.
* Hypogonadism diagnosis with not having received hormonal replacement previous to the study.
* Primary osteoporosis diagnosis.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Bone turnover markers (from baseline to 12 months under treatment) | Time frame: from baseline, 3 and 12 months under treatment.
  Plasma measure of (through LEGENDplex (Multiplex)):
  Bone formation panel that include: Osteoprotegerin (OPG) measure in pg/mL, Alkaline Phosphatase Liver/Bone/Kidney (ALPL) measure in pg/mL, LEPTINA measure in pg/mL and Bone Morphogenetic Protein 2 (BMP-2) measure in pg/mL. Bone resorption panel that include: Osteopontin (OPN) measure in pg/mL, Acid Phosphatase 5 Tartrate Resistant (ACP5) measure in pg/mL, RANKL measure in pg/mL, Tumor Necrosis Factor Alpha (TNF-α) measure in pg/mL, Interleukin 6 (IL-6) measure in pg/mL, Parathyroid Hormone (PTH) measure in pg/mL, Interleukin 1 beta (IL-1β) measure in pg/mL, Dickkopf WNT Signaling Pathway Inhibitor 1 (DKK-1) measure in pg/mL.
Change from baseline of Bone mineral density at 12 months | Time frame: from baseline and 12 months under treatment.
  Bone mineral density through Dual-energy X-ray absorptiometry (DXA scan) measure.
  Classification:
  Normal: T-score ≥ -1.0 Osteopenia: -2.5 < T-score < -1.0 Osteoporosis: T-score ≤ -2.5 Severe osteoporosis: T-score ≤ -2.5 with fragility fracture

SECONDARY OUTCOMES:
Tolerability of colaren vs standard treatment (conventional treatment): grading the severity of Adult and Pediatric Adverse Events Version 2.0 | Time frame: evaluate the tolerability from month 1, 3, 6, 9 and 12, under supplementation
  Evaluation of tolerability of Colaren and conventional treatment through the "Division of AIDS table for grading the severity of Adult and Pediatric Adverse Events Version 2.0, November 2014" Grade 1= Mild Grade 2= Moderate Grade 3= Severe Grade 4= Potentially

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wheater G, Elshahaly M, Tuck SP, Datta HK, van Laar JM. The clinical utility of bone marker measurements in osteoporosis. J Transl Med. 2013 Aug 29;11:201. doi: 10.1186/1479-5876-11-201. PMID 23984630
- [Result] Sattui SE, Saag KG. Fracture mortality: associations with epidemiology and osteoporosis treatment. Nat Rev Endocrinol. 2014 Oct;10(10):592-602. doi: 10.1038/nrendo.2014.125. Epub 2014 Aug 5. PMID 25091729
- [Result] Rothman MS, Bessesen MT. HIV infection and osteoporosis: pathophysiology, diagnosis, and treatment options. Curr Osteoporos Rep. 2012 Dec;10(4):270-7. doi: 10.1007/s11914-012-0125-0. PMID 23100110
- [Result] Panayiotopoulos A, Bhat N, Bhangoo A. Bone and vitamin D metabolism in HIV. Rev Endocr Metab Disord. 2013 Jun;14(2):119-25. doi: 10.1007/s11154-013-9246-8. PMID 23657562
- [Result] Leal J, Gray AM, Prieto-Alhambra D, Arden NK, Cooper C, Javaid MK, Judge A; REFReSH study group. Impact of hip fracture on hospital care costs: a population-based study. Osteoporos Int. 2016 Feb;27(2):549-58. doi: 10.1007/s00198-015-3277-9. Epub 2015 Aug 19. PMID 26286626
- [Result] Compston J, Cooper A, Cooper C, Gittoes N, Gregson C, Harvey N, Hope S, Kanis JA, McCloskey EV, Poole KES, Reid DM, Selby P, Thompson F, Thurston A, Vine N; National Osteoporosis Guideline Group (NOGG). UK clinical guideline for the prevention and treatment of osteoporosis. Arch Osteoporos. 2017 Dec;12(1):43. doi: 10.1007/s11657-017-0324-5. Epub 2017 Apr 19. PMID 28425085
- [Result] Bolland MJ, Grey AB, Horne AM, Briggs SE, Thomas MG, Ellis-Pegler RB, Woodhouse AF, Gamble GD, Reid IR. Annual zoledronate increases bone density in highly active antiretroviral therapy-treated human immunodeficiency virus-infected men: a randomized controlled trial. J Clin Endocrinol Metab. 2007 Apr;92(4):1283-8. doi: 10.1210/jc.2006-2216. Epub 2007 Jan 16. PMID 17227801
- [Result] Carlos F, Clark P, Maciel H, Tamayo JA. Direct costs of osteoporosis and hip fracture: an analysis for the Mexican Social Insurance Health Care System. Salud Publica Mex. 2009;51 Suppl 1:S108-13. doi: 10.1590/s0036-36342009000700014. PMID 19287884